CLINICAL TRIAL: NCT01058928
Title: Effects of Tracheal Tube Size on Pulmonary Aspiration Different Endotracheal Tube Size Influences Pulmonary Aspiration
Brief Title: Effects of Tracheal Tube Size on Pulmonary Aspiration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Jin-Young Hwang/ M.D., Seoul National University Bundang Hospital
Other Study IDs: B-0912-090-012
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2009-12

CONDITIONS: The Reduction of Aspiration Rate in Intubated Patients
Keywords: Tracheal tube; Size

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group ID 7.5: Patients with a tracheal tube ID (internal diameter) 7.5 mm
  Interventions: Other: Observation of fluid leakage around tracheal tube cuffs
- Group ID 8.0: Patients with a tracheal tube ID 8.0 mm
  Interventions: Other: Observation of fluid leakage around tracheal tube cuffs

INTERVENTIONS:
Other: Observation of fluid leakage around tracheal tube cuffs — One milliliter of Evans blue diluted in 3.5 mL of saline solution is carefully instilled on the top of the tracheal tube cuff. In the operating room, one hour and five hours after intubation, fiberoptic bronchoscopy was performed to detect the possible presence of blue dye in the trachea. If a blue spot was seen on the trachea caudal to the tube's tip on any occasion, leakage was confirmed and the experiment was finished.

SUMMARY:
Fluid leak around the cuff is minimized when the endotracheal tube size is small relative to the size of the trachea. In the current study, the investigators assess the influence of different HVLP endotracheal tube size on fluid leakage around the cuff in a benchtop model and in anesthetized patients.

DETAILED DESCRIPTION:
The use of a high-volume and low-pressure (HVLP) endotracheal cuff has reduced the cuff-induced tracheal damage because the cuff conforms passively to tracheal contours as it expands during inflation and the cuff inflation pressure is assumed to be equal to cuff-to-trachea pressure. However, longitudinal folds of a HVLP cuff occur on inflation within the trachea, as the diameter of the cuff is greater than that of the trachea, and these folds provide channels for an aspiration or gas leakage.

Silent aspiration of upper airway secretions has been reported in patients undergoing general anesthesia and in the intensive care unit (ICU). A previous study reported the 83% aspiration of subglottic dye detected by bronchoscopy in anesthetized patients, and other study of intubated patients with HVLP cuffs in the ICU showed 87% aspiration rate.

Intubation-related (ventilator associated pneumonia) pneumonia is a leading cause of prolongation of hospital stay, mortality and morbidity during the postoperative period and in the ICU. Therefore, it is important to achieve a better seal around the cuff without tracheal damage, which would reduce the incidence of pneumonia in intubated patients.

A previous benchtop study demonstrated that the leak around the cuff is minimized when the endotracheal tube size is small relative to the size of the trachea. In the current study, we assess the influence of different HVLP endotracheal tube size on fluid leakage around the cuff in a benchtop model and in anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, aged 20-65 yr scheduled for elective cardiac surgery under general anesthesia

Exclusion Criteria:

* Patients with an upper airway and vocal cord disease, pneumonia before surgery, a history of tracheostomy and tracheal stenosis.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients,scheduled for elective cardiac surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Aspiration rate | during 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Result] Pavlin EG, VanNimwegan D, Hornbein TF. Failure of a high-compliance low-pressure cuff to prevent aspiration. Anesthesiology. 1975 Feb;42(2):216-9. doi: 10.1097/00000542-197502000-00019. No abstract available. PMID 1115375
- [Result] Blunt MC, Young PJ, Patil A, Haddock A. Gel lubrication of the tracheal tube cuff reduces pulmonary aspiration. Anesthesiology. 2001 Aug;95(2):377-81. doi: 10.1097/00000542-200108000-00019. PMID 11506109